CLINICAL TRIAL: NCT02213562
Title: A Randomized, Double-blind, Parallel Group Study to Evaluate the Effect of Chrysanthemum Flower Oil and Its Dose-dependency in Subjects With Hyperuricemia
Brief Title: Effect of Chrysanthemum Flower Oil and Its Dose-dependency on Hyperuricemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: Kaneka Corporation (Industry)
Responsible Party: Principal Investigator, Fumiko Higashikawa, Associate Professor, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: eki-997
Record Dates: First submitted 2014-08-08; First posted 2014-08-11 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 200 mg CFO (Experimental): 200 mg of chrysanthemum flower oil
  Interventions: Dietary Supplement: 200 mg of chrysanthemum flower oil
- 300 mg CFO (Experimental): 300 mg of chrysanthemum flower oil
  Interventions: Dietary Supplement: 300 mg of chrysanthemum flower oil
- 400 mg CFO (Experimental): 400 mg of chrysanthemum flower oil
  Interventions: Dietary Supplement: 400 mg of chrysanthemum flower oil

INTERVENTIONS:
Dietary Supplement: 200 mg of chrysanthemum flower oil
  Arms: 200 mg CFO
Dietary Supplement: 300 mg of chrysanthemum flower oil
  Arms: 300 mg CFO
Dietary Supplement: 400 mg of chrysanthemum flower oil
  Arms: 400 mg CFO

SUMMARY:
The aim of this study is to investigate the efficacy and dose-dependency of chrysanthemum flower oil in suppressing serum uric acid.

ELIGIBILITY:
Inclusion Criteria:

* Serum uric acid 6.8-8.9 mg/dL

Exclusion Criteria:

* Taking anti-hyperuricemic drugs
* History of gouty attack
* Taking drugs or functional food that may affect serum uric acid level
* Hypertention, hyperlipidemia, or diabetes millitus
* Participation in any clinical trial within 90 days of the commencement of the trial
* Renal or hepatic dysfunction
* Heart disease
* History of severe disease and/or major surgery

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in serum uric acid from baseline | Every 4 weeks (Overall 8 weeks)
Change in uric acid clearance from baseline | Every 4 weeks (Overall 8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Fumiko Higashikawa, PhD, Principal Investigator — Hiroshima University
Locations (1):
- Hiroshima University, Hiroshima, Japan